CLINICAL TRIAL: NCT04229784
Title: Multicentrique Prospective Evaluation of Radiofrequency Surgical Treatment of Homorrhoidal Disease
Acronym: RF-GREP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr Abramowitz (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A03220-55
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-09

CONDITIONS: Hemorrhoids; Surgical Procedure, Unspecified
Keywords: hemorrhoids; radiofrequency surgery
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RF ARM (Experimental): The research procedure consists of radiofrequency destruction of hemorrhoidal vascular tissue. It consists in delivering a 4 MHz radiofrequency wave current delivered at low temperature by microfibre electrodes using a large disposable needle within the hemorrhoidal vascular tissue
  Interventions: Procedure: Radiofrewuency surgery

INTERVENTIONS:
Procedure: Radiofrewuency surgery — The research procedure consists of radiofrequency destruction of hemorrhoidal vascular tissue. It consists in delivering a 4 MHz radiofrequency wave current delivered at low temperature by microfibre electrodes using a large disposable needle within the hemorrhoidal vascular tissue

SUMMARY:
Hemorrhoids consist of a tissue rich in blood vessels and are present in all individuals inside the anus. Hemorrhoidal disease (HD) is when hemorrhoids become troublesome and cause symptoms such as pain, bleeding, prolapse or seepage.

The first steps in the treatment of HD involve either drugs or instrumental gestures (sclerosis, ligation). In the event of failure or of a disease that is significant from the outset, it is possible to envisage a surgical treatment.

The use of a radiofrequency is a new technique, already used frequently by vascular surgeons in the treatment of varicose veins of the lower limbs. This technique has been developed for radiofrequency destruction of hemorrhoidal vascular tissue.

In France, no studies have been carried out to evaluate this new technique.

DETAILED DESCRIPTION:
Hemorrhoids consist of a tissue rich in blood vessels and are present in all individuals inside the anus (internal hemorrhoids). Hemorrhoidal disease (HD) is when hemorrhoids become troublesome and cause symptoms such as pain, bleeding, prolapse or seepage.

The first steps in the treatment of HD involve either drugs or instrumental gestures (sclerosis, ligation). In the event of failure or of a disease that is significant from the outset, it is possible to envisage a surgical treatment.

The use of a radiofrequency current (Rafaelo technique) in the treatment of hemorrhoidal disease is a new technique, already used frequently by vascular surgeons in the treatment of varicose veins of the lower limbs. This technique has been developed for radiofrequency destruction of hemorrhoidal vascular tissue.

Although radiofrequency destruction of hemorrhoidal vascular tissue is already used in other European countries such as Poland, Germany, Belgium and Great Britain, there are very few studies on this minimally invasive surgical technique. This is particularly the case in France where no studies have been carried out to evaluate this new technique.

ELIGIBILITY:
Inclusion Criteria:

* Male and female consultant for a grade II or III haemorrhoidal pathology after failure of medical-instrumental treatments.
* Age > 18 years old and < 75 years old
* Patient having signed an informed consent
* Affiliate or beneficiary of a social security scheme
* For patients taking anti-vitamin K (AVK) or oral anticoagulants (OACs) a short stop will be recommended according to HAS recommendations.
* For patients on antiplatelet agents (APA), the relay and stopping procedures will be carried out according to the current recommendations of the HAS (26)
* Patient eligible to be an outpatient

Exclusion Criteria:

* Patient with IBD (inflammatory bowel diseases)
* Patient with haematological disease at risk of bleeding
* Patient with anal fistulas
* Patient unable to interrupt VKAs, OACs or APAs.
* Patient with an associated anal fissure
* External hemorrhoidal pathology
* Patient participating in another clinical study
* Pregnant or lactating women
* Patient with pacemaker or implantable defibrillator
* Protected patient: adult under guardianship, trusteeship or other legal protection, deprived of liberty by judicial or administrative decision

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
HEMO-FISS-QoL | 3 months
  The primary endpoint for assessing changes in the patient's quality of life will be the total score obtained on the HEMO-FISS-QoL Quality of Life Questionnaire at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- BLOMET clinic, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Laurain A, Bouchard D, Rouillon JM, Petit P, Liddo A, Vinson Bonnet B, Venara A, Didelot JM, Bonnaud G, Senejoux A, Higuero T, Delasalle P, Tarrerias AL, Devulder F, Castinel A, Thomas C, Pillant Le Moult H, Favreau-Weltzer C, Abramowitz L. French multicentre prospective evaluation of radiofrequency ablation in the management of haemorrhoidal disease. Tech Coloproctol. 2023 Oct;27(10):873-883. doi: 10.1007/s10151-023-02787-1. Epub 2023 Apr 2. PMID 37005961